CLINICAL TRIAL: NCT04823117
Title: The Effect of Therapeutic Use of Music on Quality of Life in Fibromyalgia Patients: a Randomized Controlled Trial
Brief Title: The Effect of Music on Quality of Life in Fibromyalgia Patients
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Cagla Ozdemir, family medicine specialist, Diskapi Teaching and Research Hospital
Other Study IDs: 34/13
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Fibromyalgia; Music Therapy; Quality of Life
Keywords: fibromyalgia; music therapy; fibromyalgia Impact Questionnaire
MeSH Terms: conditions — Fibromyalgia | interventions — Music Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Music therapy group: Music therapy lasted 30 minutes every day for a total of 20 days.
  Interventions: Other: music therapy
- Control group: No treatment given.

INTERVENTIONS:
Other: music therapy — music includes nature sounds recommended by the Turkish Psychological Association
  Groups: Music therapy group

SUMMARY:
This study's aim was to determine the effect of music therapy on symptoms and functions in patients with fibromyalgia syndrome (FMS).

DETAILED DESCRIPTION:
This study's aim was to determine the effect of music therapy on symptoms and functions in patients with fibromyalgia syndrome (FMS). Women diagnosed with FMS for at least 6 months included in the study. 16 patients were in the music treatment group and 51 patients were in the control group. Patients in music treatment group were given a music CD which includes nature sounds recommended by the Turkish Psychological Association. The patients were evaluated with Fibromyalgia Impact Questionnaire (FIQ) before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over the age of 18
* Being diagnosed as FMS according to 2010 American College of Rheumatology (ACR) criteria for FMS
* Having the diagnosis of FMS at least six months

Exclusion Criteria:

* Patients with hearing problems, pregnancy, another accompanying central sensitization syndrome or schizophrenia
* Patients with psychiatric illness
* Patients whose pharmacological treatment for FMS changed within the last three months
* Patients without a listening device
* Patients who do not have a cognitive level to answer the questions in the scale

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with fibromyalgia, admitted to polyclinics
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | 6 months
  Changes in Fibromyalgia Impact Questionnaire, the total score is between 0-100. Higher total scores indicate higher disability

CONTACTS AND LOCATIONS:
Overall Officials: Çağla Özdemir, Principal Investigator — Dışkapı Eğitim ve Araştırma Hastanesi
Locations (1):
- Çağla Özdemir, Merkez, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garza-Villarreal EA, Wilson AD, Vase L, Brattico E, Barrios FA, Jensen TS, Romero-Romo JI, Vuust P. Music reduces pain and increases functional mobility in fibromyalgia. Front Psychol. 2014 Feb 11;5:90. doi: 10.3389/fpsyg.2014.00090. eCollection 2014. PMID 24575066
- [Background] Alparslan GB, Babadag B, Ozkaraman A, Yildiz P, Musmul A, Korkmaz C. Effects of music on pain in patients with fibromyalgia. Clin Rheumatol. 2016 May;35(5):1317-21. doi: 10.1007/s10067-015-3046-3. Epub 2015 Aug 6. PMID 26245724
- [Background] Korhan EA, Uyar M, Eyigor C, Hakverdioglu Yont G, Celik S, Khorshid L. The effects of music therapy on pain in patients with neuropathic pain. Pain Manag Nurs. 2014 Mar;15(1):306-14. doi: 10.1016/j.pmn.2012.10.006. Epub 2013 Jan 31. PMID 23375348